CLINICAL TRIAL: NCT02979288
Title: Treatment of the Intermediate Vaginal Microbiota With Vaginal Probiotics Containing Lactobacillus Casei Rhamnosus (Lcr Regenerans) to Improve Pregnancy Outcomes
Brief Title: Treatment of the Intermediate Vaginal Microbiota With Vaginal Lactobacillus Casei Rhamnosus to Improve Pregnancy Outcome
Acronym: LCR35&PTD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Associate Prof. Ljubomir Petricevic MD, Associate Professor, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MUV 012017
Record Dates: First submitted 2016-11-28; First posted 2016-12-01 (Estimated); Last update posted 2021-02-24 (Actual); Status verified 2018-08

CONDITIONS: Lactobacillus Infection

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- A Nugent 4 + Lactobacilli (Experimental): Intermediate vaginal Flora Nugent 4 with Lactobacilli. Intervention with vaginal probiotics with 'Lactobacillus casei rhamnosus (Lcr 35 regenerans)
  Interventions: Drug: Lactobacillus casei rhamnosus (Lcr 35 regenerans)
- B Nugent 4 + Lactobacilli (Active Comparator): Intermediate vaginal Flora Nugent 4 with Lactobacilli, NO Intervention
  Interventions: Other: NO Intervention
- C Nugent 4 NO Lactobacilli (Experimental): Intermediate vaginal Flora Nugent 4 NO Lactobacilli, Intervention with vaginal probiotics, with 'Lactobacillus casei rhamnosus (Lcr 35 regenerans)
  Interventions: Drug: Lactobacillus casei rhamnosus (Lcr 35 regenerans)
- D Nugent 4 NO Lactobacilli (Active Comparator): Intermediate vaginal Flora Nugent 4 NO Lactobacilli, No Intervention
  Interventions: Other: NO Intervention

INTERVENTIONS:
Drug: Lactobacillus casei rhamnosus (Lcr 35 regenerans) — Probiotic vaginal tablets vith active probiotic strains
  Other Names: Gynophilus
  Arms: A Nugent 4 + Lactobacilli; C Nugent 4 NO Lactobacilli
Other: NO Intervention — NO Intervention
  Other Names: NO Medication
  Arms: B Nugent 4 + Lactobacilli; D Nugent 4 NO Lactobacilli

SUMMARY:
In the currently presented trial, investigators aim to evaluate the treatment of the intermediate vaginal microbiota during the first trimester of pregnancy with vaginal lactobacilli to restore the normal vaginal microbiota and therewith reduce the rate of PTD. All pregnant women between 10 + 0 (10 weeks plus 0 days) and 16 + 0 (16 weeks plus 0 days) gestational weeks in study group will be treated with vaginal Lactobacilli Capsules containing L. Casei rhamnosus LCR 35

DETAILED DESCRIPTION:
Despite recent achievements in perinatal care, the prevention of preterm delivery (PTD) remains a major challenge in modern obstetrics. Healthy vaginal flora, dominated by Lactobacillus species (spp.), plays an important role in the protection against genital infections, which are considered a frequent cause of PTD. Imbalances of the vaginal flora caused by a reduction in the proportion of Lactobacillus spp. can lead to an overgrowth of mixed anaerobic bacteria, which can ultimately result in bacterial vaginosis (BV). Since the effect of treating pregnant women with an abnormal vaginal flora was introduced, BV has gained interest and is now a well-known risk factor for ascending infections and subsequent PTD. However, the overall risk reduction of PTD through antibiotic treatment of an abnormal flora was disproved by large and well-designed studies in a general obstetrical population.

At present, little is known about the role of the intermediate vaginal flora, which can either be regarded as the transition from a healthy to an abnormal flora or as the transition from abnormal flora back to a healthy vaginal microbiota. The intermediate vaginal flora constitutes a highly heterogeneous group that may or may not include vaginal Lactobacillus spp. and that may or may not be characterised by the presence of anaerobic bacteria. In 2007, a meta-analysis reported that the presence of intermediate vaginal flora was not associated with PTD, late miscarriage, maternal or neonatal infection, or perinatal mortality. In contrast, an observational study by Hay et al.reported a high rate of late miscarriage (16-24 gestational weeks) in women with intermediate vaginal flora at an examination before 16 gestational weeks. Additionally, another study reported an association of PTD with partial BV, which is defined as streaks of BV flora in a smear that has areas of normal flora.

Latest research reported that there is an association between the intermediate vaginal flora and PTD. In one of our previous studies, intermediate flora was identified on the examined screening smears of 529/8421 (6.3%) women. In this group, 349/529 (66%) women had a Nugent score of 4, 94/529 (17.8%) had a Nugent score of 5, and 86/529 (16.2%) had a Nugent score of 6. In women with a Nugent score of 4, 232/349 (66.5%) women were assigned to the Lactobacilli group. The Non-Lactobacilli group consisted of 117/349 (33.5%) women with a Nugent score of 4 due to the total absence of any bacterial colonisation, including Lactobacillus spp. The preterm delivery rate was significantly lower in the Lactobacilli than in the Non-Lactobacilli group On follow-up smears, bacterial vaginosis rates were 9% in the Lactobacilli and 7.8% in the Non-Lactobacilli group. Hence, according to this retrospective study, the absence of vaginal Lactobacillus species and any bacterial colonisation increases the risks of preterm delivery and low birth weight in women with intermediate vaginal flora in early pregnancy.

In the currently presented trial, investigators aim to evaluate the treatment of the intermediate vaginal flora during the first trimester of pregnancy with vaginal lactobacilli to restore the normal vaginal microbiota and therewith reduce the rate of PTD.

At investigators Department, pregnancy care includes a prenatal consultation, where women registered for a planned delivery at our department between 10 + 0 (10 weeks plus 0 days) and 16 + 0 (16 weeks plus 0 days) gestational weeks. Women underwent routine screening for asymptomatic vaginal infections and characterization due to Nugent score. All women except those with a normal flora (Nugent score 0 to 3) will be asked to undergo a follow-up smear between 14 + 0 (14 weeks plus 0 days) and 22 + 0 (22 weeks plus 0 days) gestational weeks at our department. Vaginal smears will be obtained after vaginal fluid collection with sterile swabs from the lateral vaginal wall and posterior fornix vaginae. Both at first and control smear. All smears will be Gram-stained and microscopically analyzed by one of four biomedical laboratory assistants, specialized in gynecological cytopathology, at a laboratory that is certified according to DIN EN ISO 9001:2008. Nugent scores of 0 to 3 will be considered to indicate normal vaginal flora, 4 to 6 to indicate intermediate vaginal flora, and 7 to 10 to indicate BV.

The present study follows a prospective randomized observer-blinded mono-centric design. After obtaining the results of vaginal swab According to the Nugent scoring system, two groups will be assigned: (i) pregnant women with an intermediate vaginal flora and a Nugent score of 4 with vaginal lactobacilli (Control Group), versus (ii) pregnant women with an intermediate vaginal flora and a Nugent score of 4 without vaginal lactobacilli (Study Group).

Therapy will be assigned due to protocol. Each group will be divided in a study and control group. Patients of the study group will be treated with muco-adhesive slow release vaginal tablets containing 876,9 mg Lactobacillus casei rhamnosus (Lcr regenerans) in concentration of 107 CFU/ml (Groups A + C). The treatment duration will be 8 days with two tablets every 4th day. Patients of the control group will not undergo any treatment (Groups B + D). A vaginal control smear will be obtained 4-6 weeks following the first study visit.

The primary outcome parameter will be the recovery to the normal vaginal flora (Nugent score 0 to 3). Secondary outcome parameters will include (i) the gestational age at delivery, recorded as term delivery at or after 37 + 0 gestational weeks, (ii) the rate of PTD, defined as spontaneous delivery at or before 36 + 6 gestational weeks, due to preterm premature rupture of the membranes and/or preterm labor, (iii) neonatal birthweight, defined as a the weight at the time of delivery, and (iv) the rate of live birth, defined as the delivery or PTD of an infant that had an Apgar score at 1 minute of > 0.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women 10th to 16th Week of gestation

Exclusion Criteria:

* Vaginal Bleeding, Twins, vaginal infections, Antibiotics up to 4 weeks to randomisation

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2017-05-02 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
the recovery to the normal vaginal microbiota (Nugent score 0 to 3). | 4 Weeks

SECONDARY OUTCOMES:
the gestational age at delivery, recorded as term delivery at or after 37 + 0 gestational weeks | 9 Months

CONTACTS AND LOCATIONS:
Overall Officials: Ljubomir Petricevic, Prof, Study Chair — Medical University Vienna
Locations (1):
- Department of Obstetrics and Gynecology, Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Petricevic L, Witt A. The role of Lactobacillus casei rhamnosus Lcr35 in restoring the normal vaginal flora after antibiotic treatment of bacterial vaginosis. BJOG. 2008 Oct;115(11):1369-74. doi: 10.1111/j.1471-0528.2008.01882.x. PMID 18823487
- [Background] Kiss H, Petricevic L, Husslein P. Prospective randomised controlled trial of an infection screening programme to reduce the rate of preterm delivery. BMJ. 2004 Aug 14;329(7462):371. doi: 10.1136/bmj.38169.519653.EB. Epub 2004 Aug 4. PMID 15294856
- [Result] Farr A, Kiss H, Hagmann M, Machal S, Holzer I, Kueronya V, Husslein PW, Petricevic L. Role of Lactobacillus Species in the Intermediate Vaginal Flora in Early Pregnancy: A Retrospective Cohort Study. PLoS One. 2015 Dec 11;10(12):e0144181. doi: 10.1371/journal.pone.0144181. eCollection 2015. PMID 26658473
- [Result] Petricevic L, Domig KJ, Nierscher FJ, Sandhofer MJ, Fidesser M, Krondorfer I, Husslein P, Kneifel W, Kiss H. Characterisation of the vaginal Lactobacillus microbiota associated with preterm delivery. Sci Rep. 2014 May 30;4:5136. doi: 10.1038/srep05136. PMID 24875844